CLINICAL TRIAL: NCT06709404
Title: Telehealth Intervention to Address Distress and Financial Toxicity in the Care Partners of Patients Receiving Cytoreductive Surgery and Hyperthermic Intraperitoneal Chemotherapy
Brief Title: Telehealth Intervention for Improving Distress and Financial Toxicity in the Caregivers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00110615; P30CA012197 (NIH); WFBCCC 98522 (Other: Wake Forest Baptist Comprehensive Cancer Center)
Record Dates: First submitted 2024-11-25; First posted 2024-11-29 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Hematopoietic and Lymphatic System Neoplasm; Malignant Solid Neoplasm
MeSH Terms: interventions — Telemedicine; Practice Guidelines as Topic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Telehealth intervention) (Experimental): Participants receive telehealth navigation intervention which may consist of referral to specific resources for caregiving experience over 1 hour 1-4 weeks prior to patient's surgery.
  Interventions: Other: Telemedicine; Other: Survey administration; Other: Electronic health record review
- Group 2 (Usual Care) (Active Comparator): Participants receive standard caregiving experience on study.
  Interventions: Other: Survey administration; Other: Electronic health record review; Other: Best Practice

INTERVENTIONS:
Other: Telemedicine — Receive telehealth navigation intervention
  Arms: Group 1 (Telehealth intervention)
Other: Survey administration — Ancillary studies
Other: Electronic health record review — Ancillary studies
Other: Best Practice — Receive standard caregiving experience
  Arms: Group 2 (Usual Care)

SUMMARY:
This clinical trial assesses whether resource identification for primary caregivers can affect financial stress, quality of life, depression, and the general belief in the ability to cope with daily life. Caregivers of patients receiving cytoreductive surgery and hyperthermic intraperitoneal chemotherapy (CS+HIPEC) demonstrate that they endure high depressive symptom burdens and financial distress. Further, they experience symptom trajectories that differ from those of patients. In short, they require differential timing of supportive interventions. This study aims to reduce financial toxicity and distress levels and to increase self-efficacy, satisfaction and engagement with care. Information gathered from this study may help researchers determine whether telehealth interventions for caregivers may increase awareness of recommended resources that could be beneficial during caregivers journey.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the feasibility of a telehealth navigation intervention for CS+HIPEC caregivers.

SECONDARY OBJECTIVES:

I. To assess the efficacy of the intervention on financial distress and depression in intervention and standard of care caregivers.

II. To compare financial distress in intervention caregivers as compared to standard of care caregivers.

III. To compare satisfaction with care experiences in intervention caregivers as compared to standard of care caregivers.

IV. To compare self-efficacy for navigating treatment-related costs in intervention caregivers as compared to standard of care participants.

V. To compare self-reported community resource use among intervention and standard of care caregivers.

VI. To compare the quality of life over time in intervention caregivers as compared to standard of care caregivers.

VII. To compare social support over time in intervention caregivers as compared to standard of care caregivers.

VIII. To compare treatment satisfaction for intervention caregivers as compared to standard of care caregivers.

OUTLINE: Participants are randomized to 1 of 2 groups.

GROUP I: Participants receive telehealth navigation intervention which may consist of referral to specific resources for caregiving experience over 1 hour 1-4 weeks prior to patient's surgery.

GROUP II: Participants receive standard caregiving experience on study.

After completion of study intervention, participants are followed up at 3, 6, 12, and 24 months.

ELIGIBILITY:
Inclusion Criteria

* Primary caregiver of a patient scheduled to receive CS+HIPEC at Atrium Health Wake Forest Baptist Comprehensive Cancer Center
* Access to a computer or smartphone and must have an email address
* 18 years of age or older at the time of consent
* The ability to understand and willingness to provide written informed consent
* The ability to read and write English

Exclusion Criteria

- Patient declines access to their medical record

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01-31 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of caregivers who participate (Feasibility) | At 1 and 2 years
  Feasibility will be measured by the number of caregivers who complete the Center for Epidemiologic Studies-Depression Scale (CES-D). The 95% confidence interval for the observed rates will be calculated.

SECONDARY OUTCOMES:
Depression - Center for Epidemiologic Studies-Depression Scale (CES-D) | At pre-op, 2 weeks-3 months post-op, and 6-9 months post-op
  Depression will be based on the proportion of caregivers screening in with scores at or above 16, the score that indicates possible depression. These data will be dichotomized into depressed (yes/no) status and analyzed using a repeated measures logistic regression to see if the rate of depression changes. The model will include a time group interaction, and if that test is not significant, the term will be removed and the model refit to assess differences between groups and estimate change in CES-D score. The CES-D is a 20-item self-report measure developed to screen for depressive disorders. A score of ≥ 16 has been used as the cut-off score with higher scores indicating significant depressive symptoms. Caregivers who score ≥16 will be documented.
Financial distress - Comprehensive Score for Financial Toxicity-Functional Assessment of Chronic Illness Therapy | At pre-op, 2 weeks-3 months post-op, and 6-9 months post-op
  Will be measured using the adapted Comprehensive Score for Financial Toxicity-Functional Assessment of Chronic Illness Therapy item for caregivers. Repeated measures longitudinal models will be used to detect changes in these measures. Initially, the model will include a time group interaction, and if that test is not significant, the term will be removed and the model refit to assess differences between groups and estimate change in financial distress scores. Lower scores indicate greater financial distress; higher scores indicate better financial well being. Scores range from 0 to 44.
Satisfaction with telehealth intervention - Caregiver Reflection of Intervention Form | At post-op, at 6 months and 12 months
  The results will be summarized and reported. This item is given once to the caregivers; these results will help to make changes to the intervention in future studies. Satisfaction scores will be compared between the 2 arms using an independent t-test.
Self-efficacy | At pre-op, 2 weeks-3 months post-op, and 6-9 months post-op
  The General Self Efficacy Scale is a ten-item scale with Likert-type items created to "assess a general sense of perceived self-efficacy with the aim in mind to predict coping with daily hassles as well as adaptation after experiencing all kinds of stressful life events. Scores range from 10 to 40 with higher scores indicating greater self-efficacy
Self-reported community resource | At pre-op, 2 weeks-3 months post-op, and 6-9 months post-op
  Will be used among intervention and standard of care caregivers and will be reported as a proportion using these resources. The corresponding 95% confidence interval will also be reported. These rates can be compared between groups using a two-proportion Z-test.
Caregiver quality of life - Caregiver Quality of Life Index-Cancer (CQOLC) | At pre-op, 2 weeks, 3 months post-op, 6-9 months post-op, 12-16 months post-op, and 24-28 months post-op
  Will be measured using the Caregiver Quality of Life Index-Cancer scale for caregivers. Will be evaluated using repeated measures regression, with estimates of scores at the 5 time points reported and tested for differences across the 5 collection times. The CQOLC scale consists of 35 five-point Likert-type items. Scores range from 0-140 (Good 0-45, fair 46-90, poor 91-140). The CQOLC is made up of four subscales: Burden, Disruptiveness, Positive adaptation, and Financial concerns.
Social support - Medical Outcome Study Social Support Survey (MOS-SSS) | At pre-op, 2 weeks-3 months post-op, 6-9 months post-op, 12-16 months post-op, and 24-28 months post-op
  The MOS-SSS contains 19 functional support items hypothesized to measure five dimensions of social support: 1) emotional support, 2) informational support, 3) tangible support, 4) positive social interaction, and 5) affectionate support. Responses are on a five-point Likert-type scale ranging from 'none of the time' to 'all of the time.' Score range is 0-20. Total score is calculated by adding up the responses for each item. A higher score indicates a greater level of perceived social support.
Treatment satisfaction - Family Satisfaction with End-of-Life Care (FAMCARE) | At 2 weeks-3 months post-op and 6-9 months post-op
  The FAMCARE scale is a 20-item self-report questionnaire that measures how satisfied family caregivers are with the healthcare provided to the patient and themselves. The scale uses a Likert scale ranging from 1 to 5, with 1 being "very satisfied" and 5 being "very dissatisfied". The FAMCARE scale can be scored as mean scores or percentages. The percentage score ranges from 20 to 100, with higher scores indicating greater caregiver satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No